CLINICAL TRIAL: NCT04485260
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of KRT-232 Combined With Ruxolitinib in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera MF (Post-PV-MF), Or Post-Essential Thrombocythemia MF (Post ET-MF) Who Have a Suboptimal Response to Ruxolitinib
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-109
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Myelofibrosis
Keywords: navtemadlin
MeSH Terms: conditions — Primary Myelofibrosis | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A, Arm 1, Cohort 1 (Experimental): KRT-232 by mouth once daily for Days 1-7, off treatment for Days 8-28 (28 day cycle)
  Interventions: Drug: KRT-232; Drug: Ruxolitinib

INTERVENTIONS:
Drug: KRT-232 — administered by mouth
Drug: Ruxolitinib — administered by mouth
  Other Names: Jakafi; Jakavi

SUMMARY:
This is a phase 1b/2 study of KRT-232 combined with ruxolitinib in subjects with MF who have a suboptimal response after at least 18 weeks of treatment with ruxolitinib. The primary objective of the study is to determine a recommended phase 2 dose (RP2D) of KRT 232 in combination with ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PMF, post-PV MF, or post-ET MF, as assessed by treating physician according to the World Health Organization (WHO)
* Treatment with ruxolitinib for ≥18 weeks prior to study entry, and on a stable dose of ruxolitinib in the 8 weeks prior to study entry
* Spleen ≥5 cm palpable below the LLCM or ≥450 cm3 by MRI or CT
* Patients must have at least 2 symptoms with a score of at least 1 on the MFSAF v4.0
* ECOG performance status of 0 to 2

Exclusion Criteria:

* Patients who are positive for TP53 mutations
* Documented disease progression or clinical deterioration any time while on ruxolitinib treatment
* Patients who have had a documented spleen response to ruxolitinib.
* Prior splenectomy
* Prior MDM2 inhibitor therapy or p53-directed therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
For Phase 1: To determine the KRT-232 RP2D in combination with ruxolitinib | 15 months
  Dose limiting toxicities will be used to establish the MTD of KRT-232 in combination with ruxolitinib. Subsequently, RP2D will be based on safety and efficacy data of the combination.
For Phase 2:To determine the spleen volume reduction (SVR) at Week 24 | 6 months after last patient enrolled
  The proportion of subjects achieving SVR of ≥ 35% at Week 24 by MRI/CT scan

SECONDARY OUTCOMES:
To determine spleen response | 43 months
  The proportion of subjects achieving ≥35% SVR at any time point from Baseline while on study, as assessed by MRI (or by CT scan for applicable subjects)
To determine the change in Total Symptom Score (TSS) based Myelofibrosis Symptom Assessment Form version 4.0 (MFSAF v4.0) | 43 months
  The percentage change in TSS as measured by the MFSAF v4.0 at any time point from Baseline while on study

CONTACTS AND LOCATIONS:
Locations (38):
- United States (8):
  - City of Hope, Duarte, California
  - John Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Royal Adelaide Hospital, Adelaide, Australia
- Bulgaria (3):
  - Dr. Georgi Stranski, Pleven
  - Saint Ivan Rilski Hospital, Sofia
  - University Mutiprofile Hospital Alexandrovska, Sofia
- France (7):
  - CHU de Caen, Caen, Cedex 9
  - Chu Angers, Angers
  - Centre Hospitalier du Mans, Le Mans
  - Institut Paoli-Calmettes, Marseille
  - CHU Saint Eloi, Montpellier
  - Hopital Saint Louis, Paris
  - CHU Tours - Hôpital Bretonneau, Tours
- Germany (5):
  - Universitätsklinikum Aachen Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation, Aachen
  - Department für Innere Medizin Universitätsklinik und Poliklinik für Innere Medizin IV Hämatologie/Onkologie, Halle
  - Universitaetsklinikum Jena, Jena
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz III. Med. Klinik und Poliklinik, Mainz
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
- Shamir Medical Center ( Assaf Harofeh), Ẕerifin, Israel
- Italy (5):
  - Bologna University Hospital, Institute of Hematology, Bologna
  - Universita degli Studi di Catania, Catania
  - University of Florence, Florence
  - Istituto Tumori della Romagna (IRST), Meldola
  - Ospedale di Circolo e Fondazione MacchiASST Sette Laghi, Varese
- Poland (2):
  - Oddział Kliniczny Hematologii Szpitala Uniwersyteckiego w Krakowie, Krakow
  - Szpital Wojewódzki w Opolu Sp zooOddzial Kliniczny Hematologii, Opole
- Spain (6):
  - d'Hebron University Hospital in Barcelona, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital de Dia Quiron Zaragoza, Zaragoza